CLINICAL TRIAL: NCT06434675
Title: Anatomical Variants of Nasal Cavities and Nasal Septum in Nepalese Patients: A Retrospective Cross-Sectional Study at a Tertiary Care Center
Brief Title: Prevalence of Variants of Nasal Cavity and Nasal Septum in Nepalese
Status: Completed | Type: Observational
Sponsor: Grande International Hospital, Nepal (Other)
Responsible Party: Principal Investigator, PRAJWAL DAHAL, Principal Investigator, Grande International Hospital, Nepal
Other Study IDs: 15/2023
Record Dates: First submitted 2024-05-19; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Nasal Septum; Deviation, Congenital
Keywords: Nasal Septum; Nasal Cavity; Turbinate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Polyps: Patients evaluated for nasal polyps
  Interventions: Other: No intervention done

INTERVENTIONS:
Other: No intervention done — No intervention done

SUMMARY:
A retrospective study was conducted on 343 patients. CT PNS and head of the patients were evaluated for variants of nasal septum and nasal cavity.

DETAILED DESCRIPTION:
A retrospective study was conducted on 343 patients aged 13 years and above. Two investigators, each with 3 to 4 years of experience in the field of radiology, evaluated computed tomography scans of the paranasal sinuses and the head of these patients. The nasal septum was evaluated for degree and types of variants. Various variants of nasal cavities and nasal septum were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1)Patients undergoing NCCT PNS and Head for chronic rhinosinusitis, headache and vertigo

Exclusion Criteria:

1. Patient less than 13 years age
2. Patients with recent trauma
3. Patient with large mass/ extensive polyposis

Ages: 13 Years to 91 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient of age 13 years and more undergoing NCCT PNS and Head for chronic rhinosinusitis , headache and vertigo
Sampling Method: Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of variants of Nasal septum | 6 months
  Prevalence of deviated nasal septum will be calculated. Among those with nasal septum deviation, frequency of deviation to right, left and S shaped nasal septum will be evaluated. Nasal septal deviation angle will be measured and grading will be done.
Prevalence of variants of nasal cavity | 6 months
  Prevalence of variants of nasal cavities like hypertrophied turbinate, paradoxical turbinate, concha bullosa, lamellar concha will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: PRAJWAL DAHAL, Principal Investigator — Grande International Hospital
Locations (1):
- Prajwal Dahal, Kathmandu, Bagmati, Nepal